CLINICAL TRIAL: NCT01450371
Title: Interferential Electrical Stimulation Improves Peripheral Vasodilatation in Healthy Individuals: A Randomized Crossover Study
Brief Title: Interferential Electrical Stimulation and Vasodilatation in Healthy Individuals
Acronym: InterM
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: University of Brasilia (Other)
Responsible Party: Principal Investigator, GASPAR ROGERIO DA SILVA CHIAPPA, Principal Investigator, Gaspar Rogério da Silva Chiappa, Hospital de Clinicas de Porto Alegre
Other Study IDs: 11-0374
Record Dates: First submitted 2011-08-26; First posted 2011-10-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Decreased Vascular Flow
Keywords: Autonomic Nervous System; Neuromodulation; Blood flow control; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Interferential: The individuals are treated acutely with interferential electrical stimulation (IES) during 30 min, providing a continuous flow of symmetrical rectangular interferential current biphasic pulses using bipolar electrodes with two channels and a slope of 1/5/1. The fixed current is adjusted to 4000 Hz, with the current AMF at 100 Hz and an AMF variation of 25 Hz (25% of AMF).
  Interventions: Device: Interferential
- Placebo: The same instructions and electrode positions were provided to the placebo, although the equipment did not provide any stimulation current
  Interventions: Device: Interferential Placebo

INTERVENTIONS:
Device: Interferential — The individuals are treated acutely with IES during 30 min, providing a continuous flow of symmetrical rectangular interferential current biphasic pulses using bipolar electrodes with two channels and a slope of 1/5/1. The fixed current is adjusted to 4000 Hz, with the current AMF at 100 Hz and an AMF variation of 25 Hz (25% of AMF).
  Other Names: Transcutaenous electrical stimuation
  Groups: Interferential
Device: Interferential Placebo — The same instructions and electrode positions were provided to the placebo, although the equipment did not provide any stimulation current
  Groups: Placebo

SUMMARY:
Interferential electrical stimulation (IES) increases local blood flow. It is not known whether increases in blood flow may be caused by inhibition of sympathetic activity, mediated by muscle metaboreflex activity. The purpose of this study was to evaluate the effect of IES on metaboreflex activation in healthy subjects.

DETAILED DESCRIPTION:
The study sample consisted of 11 healthy young individuals. All subjects were non-smokers, non-obese and free of any signs or symptoms of disease, as revealed by medical history, physical examination and electrocardiogram at rest and during cardiopulmonary exercise testing. Exclusion criteria were pregnancy, breast-feeding, alcohol or drug abuse, and any medication with potential effects on cardiovascular variables. Subjects were asked not to drink caffeine-containing drinks or exercise for at least 12 and 48 hours, respectively, before the experimental protocols.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are non-smokers
* non-obese
* and free of any signs or symptoms of disease

Exclusion Criteria:

* Pregnancy
* breast-feeding
* alcohol or drug abuse
* medication with potential effects on cardiovascular variables

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects without degenerative diseases.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Muscle Metaboreflex Reflex | Participants will be followed for the duration of metaboreflex activity (up to 30 minutes)
  Calf blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Gaspar R Chiappa, Dr, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (3):
- Brazil (3):
  - University of Brasilia, Brasília, Federal District
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Gaspar Rogério da Silva Chiappa, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] Vieira PJ, Ribeiro JP, Cipriano G Jr, Umpierre D, Cahalin LP, Moraes RS, Chiappa GR. Effect of transcutaneous electrical nerve stimulation on muscle metaboreflex in healthy young and older subjects. Eur J Appl Physiol. 2012 Apr;112(4):1327-34. doi: 10.1007/s00421-011-2084-z. Epub 2011 Jul 28. PMID 21796410